CLINICAL TRIAL: NCT06050161
Title: Minimally Invasive Gynecologic Surgery Utilizing the Artisential Articulating Laparoscopic Instruments
Brief Title: Evaluating Artisential Laparoscopic Instruments in Gynecologic Surgery
Acronym: MIGS-ART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kern Medical Center (Other)
Collaborators: Livs Med (Unknown)
Responsible Party: Principal Investigator, Yufan Chen, Chief, Division of Urogynecology, Department of Obstetrics and Gynecology, Kern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KM23033
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Organ Prolapse; Abnormal Uterine Bleeding; Mesh Augmentation; Laparoscopic Surgery; Robotic Surgical Suturing; Laparoscopic Hysterectomy; Minimally Invasive Surgery
Keywords: Laparoscopic surgery; Laparoscopic suturing; Laparoscopic instruments; Pelvic organ prolapse; Sacrocolpopexy; Minimally invasive surgery; Vaginal cuff closure
MeSH Terms: conditions — Pelvic Organ Prolapse; Metrorrhagia

STUDY DESIGN:
Intervention Model Description: Those in the study scheduled for a laparoscopic hysterectomy will be randomly selected for the Artisential vs. Robotic vs. Laparoscopic vaginal cuff closure.
  Those in the study scheduled for sacrocolpopexy will have half the mesh sutured on by the primary surgical approach (robotic or laparoscopic) and the other half sutured on by the Artisential laparoscopic instrument
Who Masked: Participant
Masking Description: The patient will not be told which surgical approaches were used during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Artisential laparoscopic instrument (Experimental): Artisential laparoscopic instrument use for suturing during minimally invasive gynecologic surgery
  Interventions: Device: Articulating laparoscopic instrument; Device: Conventional laparoscopic instrument; Device: Robotic surgical instrument
- Conventional laparoscopic instrument (Active Comparator): Conventional ("straight stick") laparoscopic instrument use for suturing during minimally invasive gynecologic surgery
  Interventions: Device: Articulating laparoscopic instrument; Device: Conventional laparoscopic instrument; Device: Robotic surgical instrument
- Robotic instrument (Active Comparator): Robotic instrument use for suturing during minimally invasive gynecologic surgery
  Interventions: Device: Articulating laparoscopic instrument; Device: Conventional laparoscopic instrument; Device: Robotic surgical instrument

INTERVENTIONS:
Device: Articulating laparoscopic instrument — The Artisential articulating laparoscopic instrument will be evaluated for efficacy and safety in suturing during minimally invasive gynecologic surgery.
  Other Names: Artisential
Device: Conventional laparoscopic instrument — Conventional laparoscopic instruments will be evaluated for efficacy and safety in suturing during minimally invasive gynecologic surgery.
  Other Names: Straight stick laparoscopy
Device: Robotic surgical instrument — Robotic surgical instruments will be evaluated for efficacy and safety in suturing during minimally invasive gynecologic surgery.
  Other Names: Da Vinci Robot

SUMMARY:
This study evaluates the efficacy and safety of Artisential laparoscopic instruments in minimally invasive gynecologic surgery.

DETAILED DESCRIPTION:
The Artisential laparoscopic instrument is a novel device that allows multi-directional articulation during laparoscopic surgery. There are currently no studies evaluating the efficacy or safety of this device in minimally invasive gynecologic surgery. The investigators aim to compare the efficacy and safety of the Artisential instrument with conventional laparoscopic or robotic instruments.

Patients who are scheduled for a laparoscopic or robotic hysterectomy and/or laparoscopic or robotic sacrocolpopexy will be invited to participate in this study. During the suturing portion of the surgery (either vaginal cuff closure during a hysterectomy, or mesh attachment during a sacrocolpopexy), operating times and safety outcomes will be measured. The approach for vaginal cuff closure will be randomly selected. The approach for mesh attachment suturing will be based on the primary surgical approach (conventional laparoscopy or robotic) and compared to suturing with the Artisential and an internally controlled environment. Therefore, half of the knots placed during a case will be with the Artisential laparoscopic device, and the other half will be placed either with robotic instruments or conventional laparoscopic instruments.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for robotic or laparoscopic total hysterectomy
* Patient scheduled for robotic or laparoscopic sacrocolpopexy

Exclusion Criteria:

* Not a candidate for the above surgical procedures

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female assigned at birth with a uterus
Enrollment: 50 (Estimated)
Dates: Start 2023-09-20 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
Mesh suturing time | Intraoperative
  Time to complete 2 full knots. This includes needling times, knot tying times, and suture cutting times.
Vaginal cuff suturing time | Intraoperative
  Time to complete closure of the vaginal cuff

SECONDARY OUTCOMES:
Needling times | Intraoperative
  Time to pass needle through tissue
Knot tying times | Intraoperative
  Time to tie a surgeon's knot, followed by 2 square knots
Knot location | Intraoperative
  Anterior vs. Posterior knot location
Surgical complications | Intraoperative
  List of any complications that occurred during the use of any of the 3 instrument types (Artisential, conventional laparoscopic, robotic)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Darwich I, Abuassi M, Weiss C, Stephan D, Willeke F. The Artisential(R) Articulated Laparoscopic Forceps: A Dry Lab Study to Examine Dexterity and Learning Effects in Operators with Different Levels of Laparoscopic Experience. Surg Technol Int. 2021 May 20;38:29-36. doi: 10.52198/21.STI.38.SO1424. PMID 33755941
- [Background] Jung Y, Hong JI, Han KN, Kim HK. Thoracoscopic anterior mediastinal mass removal using an articulating laparoscopic instrument. Interact Cardiovasc Thorac Surg. 2021 Aug 18;33(3):498. doi: 10.1093/icvts/ivab110. No abstract available. PMID 33880541
- [Background] Kim A, Lee CM, Park S. Is it Beneficial to Utilize an Articulating Instrument in Single-Port Laparoscopic Gastrectomy? J Gastric Cancer. 2021 Mar;21(1):38-48. doi: 10.5230/jgc.2021.21.e2. Epub 2021 Mar 11. PMID 33854812
- [Background] Darwich I, Scheidt M, Koliesnikov Y, Willeke F. Laparoscopic low anterior resection performed using ArtiSential(R) in an obese male patient with a narrow pelvis - a video vignette. Colorectal Dis. 2021 Mar;23(3):757-758. doi: 10.1111/codi.15473. Epub 2020 Dec 18. No abstract available. PMID 33275820
- [Background] Trevis J, Chilvers N, Freystaetter K, Dunning J. Surgeon-Powered Robotics in Thoracic Surgery; An Era of Surgical Innovation and Its Benefits for the Patient and Beyond. Front Surg. 2020 Nov 26;7:589565. doi: 10.3389/fsurg.2020.589565. eCollection 2020. PMID 33330607
- [Background] Kang SH, Won Y, Lee K, Youn SI, Min SH, Park YS, Ahn SH, Kim HH. Single-Incision Proximal Gastrectomy With Double-Flap Esophagogastrostomy Using Novel Laparoscopic Instruments. Surg Innov. 2021 Feb;28(1):151-154. doi: 10.1177/1553350620958237. Epub 2020 Sep 16. PMID 32938322
- [Background] Jin HY, Lee CS, Lee YS. Laparoscopic extended right hemicolectomy with D3 lymph node dissection using a new articulating instrument. Tech Coloproctol. 2021 Feb;25(2):235-237. doi: 10.1007/s10151-020-02345-z. Epub 2020 Sep 14. No abstract available. PMID 32926244
- [Background] Min SH, Cho YS, Park K, Lee Y, Park YS, Ahn SH, Park DJ, Kim HH. Multi-DOF (Degree of Freedom) Articulating Laparoscopic Instrument is an Effective Device in Performing Challenging Sutures. J Minim Invasive Surg. 2019 Dec 15;22(4):157-163. doi: 10.7602/jmis.2019.22.4.157. PMID 35601367
- [Background] Lee CS, Lee YS. Laparoscopic low anterior resection using new articulating instruments. Tech Coloproctol. 2021 Nov;25(11):1259-1261. doi: 10.1007/s10151-021-02486-9. Epub 2021 Jun 17. No abstract available. PMID 34142257
- [Background] Kang SH, Cho YS, Min SH, Park YS, Ahn SH, Do Park J, Kim HH. Intracorporeal overlap gastro-gastrostomy for solo single-incision pylorus-preserving gastrectomy in early gastric cancer. Surg Today. 2019 Dec;49(12):1074-1079. doi: 10.1007/s00595-019-01820-x. Epub 2019 May 21. PMID 31115696
- [Background] Dunning J. Disruptive technology will transform what we think of as robotic surgery in under ten years. Ann Cardiothorac Surg. 2019 Mar;8(2):274-278. doi: 10.21037/acs.2019.03.02. PMID 31032213
- [Background] Jin HY, Lee CS, Lee YS. Single Incision Laparoscopic Appendectomy Using a New Multi-joint Articulating Instrument. J Gastrointest Surg. 2021 Sep;25(9):2437-2438. doi: 10.1007/s11605-021-05026-w. Epub 2021 May 19. No abstract available. PMID 34013483
- [Background] Parente G, Thomas E, Cravano S, Di Mitri M, Vastano M, Gargano T, Cerasoli T, Ruspi F, Libri M, Lima M. ArtiSential(R) Articulated Wrist-Like Instruments and Their First Application in Pediatric Minimally Invasive Surgery: Case Reports and Literature Review of the Most Commonly Available Robot-Inspired Devices. Children (Basel). 2021 Jul 17;8(7):603. doi: 10.3390/children8070603. PMID 34356582
- [Background] Lee E, Lee K, Kang SH, Lee S, Won Y, Park YS, Ahn SH, Suh YS, Kim HH. Usefulness of articulating laparoscopic instruments during laparoscopic gastrectomy for gastric adenocarcinoma. J Minim Invasive Surg. 2021 Mar 15;24(1):35-42. doi: 10.7602/jmis.2021.24.1.35. PMID 35601278